CLINICAL TRIAL: NCT02051725
Title: Implementation of an "Active Life-style" Intervention in Older People With Low Physical Function: Effect on Functional Impairments, Pilot
Brief Title: Functional Impairments and Exercise in Older Adults With Low Physical Function,
Acronym: HANC-Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: European Union (Other); Odense University Hospital (Other); University of Pittsburgh (Other); National Institute on Aging (NIA) (NIH); Maastricht University (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Paolo Caserotti, Assistant Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HANC 104-1.5-11
Record Dates: First submitted 2014-01-03; First posted 2014-01-31 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Functionally Impaired Elderly; Aging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active life-style intervention (Experimental): The "active life-style intervention" is designed as 12-week structured and progressive heavy-resistance power training combined with recommended everyday physical activity.
  Interventions: Other: Active life-style intervention
- Control (No Intervention): The control group is offered to enroll in the same active life-style intervention after the end of the 12-week control period. During the control period this group is asked to maintain the habitual life style.

INTERVENTIONS:
Other: Active life-style intervention
  Arms: Active life-style intervention

SUMMARY:
* Aging is associated with a progressive and generalized deterioration of physiologic systems and greater incidence of chronic conditions, which ultimately translates into functional impairment, disability and dependency.
* Physical activity and exercise have been recognized as key pillars for the management of chronic diseases in support of medical treatment, and essential to increase physiologic function, but there is only limited evidence indicating increased physical function, following exercise interventions. One of the greatest challenges in the science of aging and exercise is to understand whether and to which extent exercise and active life-style may postpone the onset of disability and/or reverse physical impairments.
* Maintenance/improvements of physical function and mobility should be considered as primary targets for independent living, active engagement in societal challenges, and, more in general, when promoting "active ageing".
* The aim of this study is to collect preliminary data to identify the feasibility and sustainability of an "active life-style intervention" in older adults with reduced mobility receiving a preventive home visit from the public health care authority.
* This study will represent the base for a larger phase III parallel group study implemented in the public health care setting, with the specific aim of improving physical function and delay the onset of functional impairment in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Older adults (age 76 years and above) receiving a visit from the personnel of preventive home unit of municipality of Odense (DK)
* Mini Mental State Examination > = 21
* Self-selected gait speed < 0,9 m/s
* Ability to self-transport to the training facility

Exclusion Criteria:

* Unstable medical conditions including ECG abnormalities, uncontrolled hypertension, terminal and critical chronic conditions (e.g. cancer, severe heart failure)
* Amputation or other severe physical impairments prohibiting participation in the active life-style intervention
* Refusal to wear accelerometer

Min Age: 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Changes in leg press muscle power | Changes in muscle power from baseline to 12-week follow up
  Muscle power will be assessed on the dominant leg with the Notthingham power rig and expressed as Watt/kg. Subjects are sitting with

SECONDARY OUTCOMES:
Physical activity, sedentary behaviour and sleep quality (objectively assessed by accelerometry) | Changes from baseline to 12-week follow up
Cognitive function (Mini Mental State Examination and Digit Symbol Substitution Test) | Changes from baseline to 12-week follow up
Self-report Health-related measures including quality of life, pain, depression, sleep quality, fatigue, activities of daily living, anxiety. | Changes from baseline to 12-week follow up
Body composition including muscle, fat and bone quantity and quality | Changes from baseline to 12-week follow up
Neuromuscular function including strength, power, explosive force, postural control, motor/sensor nerve function | Changes from baseline to 12-week follow up
Selected blood biomarkers related to physical, muscle-skeletal and cognitive function (e.g. C reactive protein, insulin like growth factor, IL-6, BDNF) | Changes from baseline to 12-week follow up
Physical function including short and long distance walking speed, stair climbing, Short Physical Performance Battery Test | Changes from baseline to 12-week follow up

OTHER OUTCOMES:
Use of public health care resources | 5-year retrospectively and 3-year prospectively

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Caserotti, PhD, Principal Investigator — Department of Sports Science and Clinical Biomechanics, University of Southern Denmark
Locations (1):
- University of Southern Denmark, Department of Sports Science and Clinical Biomechanics, Odense, Denmark

REFERENCES:
- [Derived] Muollo V, Hvid LG, Shanbhogue VV, Steinhauser V, Caporossi D, Dimauro I, Andersen MS, Fantini C, Grazioli E, Strotmeyer ES, Caserotti P. Effects of 12-week power training on bone in mobility-limited older adults: randomised controlled trial. Arch Osteoporos. 2024 Dec 27;20(1):5. doi: 10.1007/s11657-024-01487-z. PMID 39729186